CLINICAL TRIAL: NCT04622761
Title: Phase II Study of the Use of Neoadjuvant Cabazitaxel With Hormonal Treatment in Patients With High Risk Operable Prostate Cancer, to Assess the Efficacy and Toxicity of Cabazitaxel, and, to Explore Potential Predictive and Prognostic Markers of Clinical Outcome
Brief Title: Phase II Study of the Use of Neoadjuvant Cabazitaxel With Hormonal Treatment in Patients Operable Prostate Cancer, Assess the Efficacy and Toxicity of Cabazitaxel, and Explore Potential Predictive and Prognostic Markers of Clinical Outcome
Acronym: CHROME
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDD630
Record Dates: First submitted 2020-09-29; First posted 2020-11-10 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; XRP6258

STUDY DESIGN:
Intervention Model Description: A two arm, phase II randomised multi-centre trial. 120 patients will be recruited to the trial. Patients will be randomised to a control arm of immediate surgery or a treatment arm in a ratio of 1:2 (control 40pts: treatment 80pts). Patients in the treatment arm will receive hormonal treatment and Cabazitaxel 25 mg/m2 day 1 intravenously over one hour every 21 days. Treatment will be continued for 4 cycles (3 months) unless disease progression, unacceptable toxicity or patient request.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): Immediate surgery (radical prostatectomy) (standard care)
- treatment (Experimental): 14 days prior to starting Cabazitaxel patients will take 50mg Bicalutamide once daily for 21 days.
  7 days prior to starting Cabazitaxel patients will be given 3 months LHRH treatment via injection. The entire dose will be administered via one injection 7 days prior to starting Cabazitaxel. This may be either leuprorelin or goserelin acetate and should be given as per local practice.
  At least 30 minutes prior to each administration of Cabazitaxel, patients will be administered IV premedication consisting of:
  50mg Ranitidine 10mg Chlorphenamine 8mg Dexamethasone Daily from Day 1 until end of Cabazitaxel treatment patients will take 10mg Prednisolone once daily from Day 1 until end of Cabazitaxel treatment Day 1 of each cycle - Patients will receive Cabazitaxel 25 mg/m2 intravenously over one hour every 21 days (on Day 1 of each cycle). Treatment will be continued for 4 cycles.
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — Patients will receive Cabazitaxel 25 mg/m2 * intravenously over one hour every 21 days (on Day 1 of each cycle). Treatment will be continued for 4 cycles unless disease progression, unacceptable toxicity or patient request. These patients will have surgery (radical prostatectomy) 4-86 weeks following treatment.
  *Cabazitaxel dose should be capped at 50mg (BSA=2)
  Other Names: jevtana, XRP6258, RPR116258A
  Arms: treatment

SUMMARY:
This study is evaluating the efficacy of cabazitaxel and hormonal treatment as neoadjuvant treatment for patients with clinically operable disease suitable for surgery, and a high risk of relapse after surgery

DETAILED DESCRIPTION:
This study is evaluating the efficacy of cabazitaxel and hormonal treatment (LHRH analogues) as neoadjuvant treatment for patients with clinically operable disease suitable for surgery (no lymph node, visceral or bony metastases), and a high risk of relapse after surgery (5 year risk of relapse).

Patients will receive four cycles of neoadjuvant treatment (cabazitaxel treatment and 3 months LHRH treatment) unless there is evidence of disease progression, unacceptable toxicity or patient request to withdraw consent.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years
2. ECOG performance status 0-1 (Appendix 2)
3. Diagnosis of high risk prostate cancer as defined by one or more of the following: clinically T2c/T3, Gleason 8-10 and or PSA >10ng/ml
4. Appropriate candidate for radical prostatectomy
5. Life expectancy greater than 10 years
6. Adequate organ function as evidenced by peripheral blood counts and serum chemistries at enrolment
7. Ability and capacity to consent and comply with study and follow-up procedures
8. Fit to receive chemotherapy

Exclusion Criteria:

1. Locally advanced or metastatic disease
2. Patients with a history of other previous malignancy except treated CIN or non melanomatous skin cancer
3. Grade ≥2 peripheral neuropathy
4. Grade ≥2 stomatitis
5. History of severe hypersensitivity reaction (≥ grade 3) to taxane
6. History of severe hypersensitivity reaction (≥ grade 3) to polysorbate 80 containing drugs
7. Other concurrent serious illness or medical conditions
8. Inadequate organ and bone marrow function as evidenced by:

   1. Haemoglobin <10.0 g/dL
   2. Absolute neutrophil count <1.5 x 109/L
   3. Platelet count <100 x 109/L
   4. AST/SGOT and/or ALT/SGPT >1.5 xULN
   5. Total bilirubin >1.5 x ULN
   6. Serum creatinine >1.5 x ULN (if creatinine is 1.0 - 1.5 xULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance <60mL/min should be excluded - see Appendix 3)
9. Uncontrolled diabetes mellitus
10. Active uncontrolled gastro oesophageal reflux disease (GORD)
11. Active infection requiring systemic antibiotic or antifungal medication
12. Participation in another clinical trial with any investigational drug within 30 days prior to study enrolment
13. Concurrent or planned treatment with strong inhibitors of cytochrome P450 3A4/5 (a 1-week washout period is necessary for patients who are already on these treatments - see Appendix 5 for a list of CYP3A inhibitors)
14. Concurrent or planned treatment with strong inducers of cytochrome P450 3A4/5 (a 1-week washout period is necessary for patients who are already on these treatments) - see Appendix 4 for a list of CYP3A inducers)
15. Contraindications or sensitivity to GCSF treatments
16. History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade > 2 (NCI CTCAE, version 4.03), thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (e.g., pericardial effusion restrictive cardiomyopathy) within 6 months prior to first dose of study drug. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2025-11-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy activity of neoadjuvant Cabazitaxel chemotherapy and hormonal therapy in patients with high risk operable prostate cancer, measuring the reduction in treatment failure and comparing this to that obtained in the control arm | through study completion, average 3 years
  Treatment failure is defined as: PSA level ≥ 0.12ng/ml measured on at least two occasions (1 confirmatory sample) post-surgery within three years of follow-up or death related to prostate cancer or use of a salvage therapy or not undergoing surgery at all.)

SECONDARY OUTCOMES:
• To assess the efficacy of neoadjuvant Cabazitaxel chemotherapy and hormonal therapy, measuring the pathological and radiological response rates and comparing this to that obtained in a control arm of immediate surgery. | 3 year follow up
  Pathological response rate assessed as per pTNM staging system Radiological response rates as defined in RECIST V1.1 Combined to give overall response rate
To assess the efficacy of neoadjuvant Cabazitaxel chemotherapy and hormonal therapy, assessing surgical margin involvement and comparing this to that obtained in a control arm of immediate surgery. | 3 year follow up
  The proportion of patients with positive resection margin will be reported and compared across the treatment groups using Chi-square tests. Multivariable models using logistic regression techniques shall be used to adjust for key prognostic variables of interest.
To assess the efficacy of neoadjuvant Cabazitaxel chemotherapy and hormonal therapy, assessing lymph node involvement and comparing this to that obtained in a control arm of immediate surgery. | 3 year follow up
  The proportion of patients with positive lymph nodes will be reported and compared across the treatment groups using Chi-square tests.
To assess the efficacy of neoadjuvant Cabazitaxel chemotherapy and hormonal therapy, measuring progression free survival and comparing this to that obtained in a control arm of immediate surgery. | 3 year follow up
• To assess the efficacy of neoadjuvant Cabazitaxel chemotherapy and hormonal therapy, measuring overall survival from time of randomisation to death and comparing this to that obtained in a control arm of immediate surgery. | 3 year follow up
To assess the efficacy of neoadjuvant Cabazitaxel chemotherapy and hormonal therapy, measuring surgical feasibility and comparing this to that obtained in a control arm of immediate surgery. | 3 year follow up
  The proportion of patients with delays to surgery, perioperative morbidities, mortalities and surgical complications will be reported and compared across the treatment groups.
To assess the quality of life of patients receiving neoadjuvant Cabazitaxel chemotherapy and hormonal therapy and comparing this to quality of life patients in a control arm of immediate surgery using the EORTC QLQ-C30 version 3 questionnaire. | 3 year follow up
  Responses to EORTC QLQ-C30 will be reported (median, IQR) according to global health status, the functional scales and symptom scales, by intervention group, and over time. Joint modelling or quality-adjusted survival analysis will be undertaken to allow a simultaneous assessment of quality of life and survival.

IPD SHARING:
Plan to Share IPD: Undecided